



## COVER PAGE

## Mind over Cervix: Using Virtual Reality to reduce Colposcopy Anxiety

VR as a distraction technique for management of acute anxiety and pain during outpatient colposcopy procedures – a single centre randomised control trial

Clincal Trials ID: FCNUR-23-098

NCT: Not yet assigned

IRAS ID: 335105

Document date and version: v2 29.12.23

REC reference: FCNUR-23-098









## PARTICIPANT CONSENT FORM

## Mind over Cervix: Using Virtual Reality to reduce Colposcopy Anxiety

| Participant Identification Number: |
|---|
| irtual Reality in Outpatient Colposcopy: A novel method of reducing patient anxiety and pain scores |

Name of Principle Researcher: Dr Victoria Braden

Please initial boxes

| 1 | I confirm I have read and understood the patient information sheet (date / version number) about the procedures and purpose of Virtual Reality in colposcopy and what my involvement will be. |
|---|---|
| 2 | I have had the opportunity to ask questions and the researcher has answered my questions to my satisfaction |
| 3 | I understand that my participation is voluntary and I am free to withdraw from the study at any time without giving any reason, without my medical care or legal rights being affected |
| 4 | I understand that my involvement in this study will involve me completing a questionnaire prior my procedure, receiving the colposcopy with or without the Virtual Reality headset, and completing a post procedure questionnaire |
| 5 | I understand and give permission that relevant parts of my medical notes may be looked at by medical researchers as part of the project. I give permission that the anonymised data taken can be stored for use in future research into colposcopy |
| 6 | I agree to take part in the above study. |

Participant Consent Form version 2 29.12.24

IRAS project ID: 335105 REC reference: FCNUR-23-098





| Name of patient | Date | Signature |
|-------------------------------|------|-----------|
| Name of person taking consent | Date | Signature |

When complete: one copy for patient, one for researcher site file, one (original) to be kept in medical notes.

If you have any queries, please do not hesitate to contact the Chief Investigator:

Claire McFeeters
Lecturer, School of Health Sciences
Ulster University
028 7167 5945 / 5942
c.mcfeeters@ulster.ac.uk

REC reference: FCNUR-23-098